CLINICAL TRIAL: NCT01292954
Title: Effects of Blueberries on Vascular Function and Blood Pressure in Healthy Men
Brief Title: Effect of Blueberries on Vascular Function in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Alpro Foundation (Other); Wild Blueberry Association of North America (Other)
Responsible Party: Dr Jeremy Spencer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UReading-2-2011
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: blueberries; vascular function; FMD; Blood pressure; Laser Doppler; pharmacokinetics; absorption; metabolism; polyphenols; flavonoids
MeSH Terms: interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose blueberry (Active Comparator)
  Interventions: Dietary Supplement: Blueberries
- medium dose blueberry (Active Comparator)
  Interventions: Dietary Supplement: Blueberries
- high dose blueberry (Active Comparator)
  Interventions: Dietary Supplement: Blueberries
- control (Placebo Comparator)
  Interventions: Dietary Supplement: Blueberries

INTERVENTIONS:
Dietary Supplement: Blueberries — low dose: 31.4 g of freeze dried blueberry reconstituted in water medium dose: 57 g of freeze dried blueberry reconstituted in water high dose: 80 g of freeze dried blueberry reconstituted in water Placebo: sugars and vitamin c match control in water Frequency:1 single time Total Duration: 3 days study over 3 weeks period

SUMMARY:
Scientific question to be addressed: To determine the effects of acute blueberry ingestion on vascular function and blood pressure in humans

Hypothesis: Acute consumption of blueberry induces an improvement in blood pressure and vascular function through the impact of blueberry flavonoids on the vascular system.

Study objectives: To determine the dose-dependency of a blueberry drink on blood pressure and vascular function in healthy subjects and to determine pharmacokinetics of blueberry polyphenols

DETAILED DESCRIPTION:
Coronary heart disease (CHD) remains one of the major causes of premature death in the world. There is now substantial evidence to indicate that the cells lining the inner surface of arteries play a major role in protection against the development and progression of CHD. This layer of cells is termed the endothelium and regulates vascular tone by promoting the expansion and contraction of the blood vessel. There are a variety of non-invasive techniques for measuring endothelial function.

Research provides evidence that consumption of a diet high in plant foods and rich in polyphenols is associated with a reduction in incidence of coronary heart disease (CHD). Polyphenols, of which the flavonoids are the largest group, are thought to play a role in the reduction of incidence of chronic diseases such as cardiovascular disease and stroke. Recent studies in humans show that flavonoid-rich foods improve peripheral blood flow and surrogate markers of cardiovascular function. These effects were associated with acute elevations in the levels of circulating nitric oxide species, an enhanced flow mediated dilatation (FMD) response of conduit arteries, and an augmented microcirculation. Increases in circulating nitric oxide species in response to flavonoid ingestion suggest that circulating flavonoids (and/or their metabolic forms) may exert positive effects on vascular tone.

The purpose of this study is to assess the impact of acute flavonoid intake on postprandial vascular reactivity of healthy volunteers. Specifically, the investigators plan to perform a randomised, double blind, cross-over human intervention trial using a blueberry drink to investigate the dose-dependent effects of blueberries using a range of techniques to measure endothelial function. The study will not only measure the acute effects of flavonoid ingestion on vascular reactivity but will also assess flavonoid and metabolite levels in blood and urine and other endothelial markers.

ELIGIBILITY:
Inclusion Criteria:

* Male
* A signed consent form
* Age 19-40 years old
* Body mass index - 18.5-30 kg/m2

Exclusion Criteria:

* Blood pressure > 150/90 mmHg
* Haemoglobin (anaemia marker) < 125 g/l
* Gamma GT (liver enzymes) > 80 IU/l
* Cholesterol > 6.5 mmol/l
* Had suffered a myocardial infarction or stroke in the previous 12 months
* Suffers from any reproductive disorder
* Suffers from any blood-clotting disorder
* Suffers from any metabolic disorders (e.g. diabetes or any other endocrine or liver diseases)
* Any dietary restrictions or on a weight reducing diet
* Drinking more than 21 units per week
* On any medication affecting blood clotting
* On any vitamin supplements/fish oil capsules
* Smoking
* Vegetarians or vegans

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | 0-6 hours after consumption

SECONDARY OUTCOMES:
Blueberry polyphenols pharmacokinetics | 0- 24 h after consumption
Blood Pressure | 0-6 hours after consumption
Laser Doppler Iontophoresis | 0-6 hours after consumption

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Rodriguez-Mateos A, Rendeiro C, Bergillos-Meca T, Tabatabaee S, George TW, Heiss C, Spencer JP. Intake and time dependence of blueberry flavonoid-induced improvements in vascular function: a randomized, controlled, double-blind, crossover intervention study with mechanistic insights into biological activity. Am J Clin Nutr. 2013 Nov;98(5):1179-91. doi: 10.3945/ajcn.113.066639. Epub 2013 Sep 4. PMID 24004888